CLINICAL TRIAL: NCT06981871
Title: Prevalence of Lower and Upper Incisor Periodontal Phenotypes and Risk Indicators in French Dental Students: a Bicentric Cross-sectional Study
Brief Title: Prevalence of Lower and Upper Incisor Periodontal Phenotypes and Risk Indicators.
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Odonto02
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Gingiva; Phenotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of the gingival phenotype of the incisors in the upper and lower jaws — Assessment of gingival thickness (Kan et al 2015) and keratinised tissue height of the incisors with UNC-15 peridontal probe (Hu-Freidy, USA) and clinical photography.

SUMMARY:
The determination of the periodontal phenotype is an essential part of the periodontal diagnostic process, which must guide not only treatment but also prognosis (Kim et al. 2020).

This determination is based on the clinical assessment of 3 individual variables: gingival height/thickness and alveolar bone cortical thickness. Although these anatomical characteristics are genetically determined, they are also influenced by numerous acquired, endogenous or exogenous factors that can act at a general and/or local level. The periodontal phenotype is therefore specific to an individual and its 3 components vary over time according to the dental sectors and sites of each individual. For example, the morphology of this phenotype varies according to whether the gingiva is thick or thin, high or reduced, and the bone cortex is thick or thin, with all possible combinations. Clinicians need to know the distribution of these different types of phenotypes, particularly in the aesthetic areas they are concerned with, in order to better identify the most fragile ones in the face of the multiple daily stresses to which the periodontium may be subjected: muscular force, dental plaque, oral hygiene manoeuvres, parafunctionality, dental procedures....

However, studies on the prevalence of the periodontal phenotype are limited and mainly concern Asian, Indian and American populations, with very few studies on European populations. Main objective: To assess the prevalence of periodontal phenotypes in the upper and lower incisors of French subjects, according to tooth type and at the individual level. Secondary objective: Identification of potential risk indicators in relation to the type of periodontal phenotype."

ELIGIBILITY:
Inclusion Criteria:

* Age (18 years old or older),
* Dental student on the university hospitals of Nice and Nancy.
* Social security affiliate.
* Systemically healthy.
* Healthy and intact periodontium.
* Informed consent.

Exclusion Criteria:

* Pregnancy.
* Under any regular medical treatment.
* Active periodontal disease.
* Enduring orthodontic treatment.
* Periodontal surgery in the mandibulary anterior region.
* Non consent patient.
* Patient under judgment trials.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Dental students at the university hospitals of Nice and Nancy (France)
Sampling Method: Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of gingival phenotypes (gingival thickness ) | At the inclusion
  Assessment of gingival thickness
Prevalence of gingival phenotypes (keratinised tissue height) | At the inclusion
  Evaluation of keratinised tissue height of the lower and upper incisors with UNC-15 peridontal probe (mm) and clinical photography.
Prevalence of gingival phenotypes (Photography) | At the inclusion
  Description of the gingiva

SECONDARY OUTCOMES:
Associated risk indicators for thin gingival phenotype ( Clinical description) | At the inclusion
  Global description clinical multiples evaluations ( Age, gender, smoking habit, orthodontic background, oral hygiene habit, oral ventilation, dysfunction, facial typology, chin shape, visibility of vascularisation and root convexity through the gum, gingival récession (Cairo), freinal insertion and skin type).
Associated risk indicators for thin gingival phenotype ( orthodontic and facial characteristics ) | At the inclusion
  Global description clinical evaluation based on photographs.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France